CLINICAL TRIAL: NCT02000856
Title: BEET PAH: a Study to Assess the Effects of Beetroot Juice in Patients With Pulmonary Arterial Hypertension
Acronym: BEET-PAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEET-PAH
Record Dates: First submitted 2013-11-19; First posted 2013-12-04 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Active Comparator): Eligible subjects will be randomised, in a double-blind crossover design, to receive treatment with either nitrate rich beetroot juice (70 ml containing approximately 8 mmol nitrate - active comparator) or nitrate depleted beetroot juice (70 ml - placebo) twice daily for 7 days (treatment period 1) followed by a 7 day washout period followed by treatment twice daily with the active comparator or placebo depending on initial treatment for another 7 days (treatment period 2) .
  Interventions: Dietary Supplement: Beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator): Eligible subjects will be randomised, in a double-blind crossover design, to receive treatment with either nitrate rich beetroot juice (70 ml containing approximately 8 mmol nitrate - active comparator) or nitrate depleted beetroot juice (70 ml - placebo)twice daily for 7 days (treatment period 1) followed by a 7 day washout period followed by treatment twice daily with the active comparator or placebo depending on initial treatment for another 7 days (treatment period 2) .
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice

SUMMARY:
The study is a single center randomised, double-blind, placebo-controlled crossover study to assess the effects of beetroot juice in patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* PAH (pulmonary arterial hypertension)
* WHO functional class II-III

Exclusion Criteria:

* WHO functional class I or IV
* pregnancy
* known intolerance or allergy to beetroot
* treatment with Allopurinol
* treatment with Iloprost (inhaled)
* systolic bloodpressure < 95 mmHg
* diabetes mellitus type 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in VO2 submax and or VO2 max | 7 days

SECONDARY OUTCOMES:
Change in 6MWT | 7 days
Change in WHO functional class | 7 days
Change in echocardiographic parameters | 7 days
  Change in; pulmonary artery systolic pressure (PASP), ventricular diastolic function, systolic right and left ventricular function, right and left atrial/ventricular dimensions will be calculated
Change in exhaled NO | 7 days
Change in systemic bloodpressure | 7 days
Change in metabolic pathways involved in nitric oxide production and regulation | 7 days
  Change in the following biochemical variables will be calculated; ADMA, SDMA, Arginine, Citrulline, Ornithine, uric acid, nitrate, nitrite
Change in NT-pro-BNP | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Wikström, MD, PhD, Principal Investigator — Uppsala University and Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden